CLINICAL TRIAL: NCT02218905
Title: Phase 0 Study of Reference Values for One Minute Sit to Stand Test in Healthy Indian Population - a Cross Sectional Study
Brief Title: Normative Values and Forming Regression Equations for One Minute Sit to Stand Test in Healthy Normal Indian Population
Acronym: 1minSTS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Baskaran Chandrasekaran (Other)
Collaborators: PSG Hospitals (Other)
Responsible Party: Sponsor-Investigator, Baskaran Chandrasekaran, Senior Physiotherapist, PSG Hospitals
Organization: PSG Hospitals (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13/311
Record Dates: First submitted 2014-08-12; First posted 2014-08-18 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Human Healthy Volunteers
Keywords: Correlation; Sit to stand repetitions; Anthropometric variables; Age; Height; weight; Gender; Regression
MeSH Terms: conditions — Body Weight; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sit to stand test (Experimental): One minute sit to stand in 40 inches armless chair. Fatigue, breathlessness and failure to maintain tempo will lead to decease the test
  Interventions: Behavioral: Sit to stand test

INTERVENTIONS:
Behavioral: Sit to stand test — Subjects will be asked to sit to stand in 40 inches chair for 60 seconds.

SUMMARY:
This study is to find relation between number of repetitions the volunteer able to sit and stand in an armless chair and their age, height, weight and gender. The investigators hypothesis there is a moderate relation between anthropometric characteristics and number of situps. This may partially define the ability of functional capacity and quadriceps ability.

DETAILED DESCRIPTION:
Sit to stand is gaining importance as a functional capacity measurement tool in modern chronic diseases arena. Bu the reference values for normative population is not available. Hence the present study aimed at finding relation between the anthropometric variables (age, height, weight) and number of sit to stand repetitions. The volunteers will be asked to sit to stand in an arm less chair of 40 inches height. The number of repetition will be correlated and regression equations will be sought out relating number of repetitions and anthropometric variables through best fit regression equations

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* 30 - 80 years old
* Hospital staffs, relatives of patients volunteering the test
* Willing to give consent for the test

Exclusion Criteria:

* Chronic cardiovascular and pulmonary diseases
* On anticoagulants
* Cancer undergoing chemo, radiotherapy
* recent orthopaedic ailments (Osteoarthritis, Rheumatoid arthritis, surgeries less than 3 months)
* Balance impairments

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Number of repetitions of sit ups within 60 seconds | baseline, 1.5 minutes

SECONDARY OUTCOMES:
heart rate recovery (in seconds) | 1 minute
blood pressure (mmHg) | baseline, 1 minute
saturation (%) | baseline, 0.5 minute, 1 minute
Heart rate (beats/ min) | baseline, 0.5 minute, 1 minute

OTHER OUTCOMES:
Anthropometric variables | Baseline
  Age, height, weight of the volunteers

CONTACTS AND LOCATIONS:
Overall Officials: RM PL Ramanathan, MD DM, Principal Investigator — PSG Hospitals
Locations (1):
- PSG Hospitals, Coimbatore, Tamil Nadu, India